CLINICAL TRIAL: NCT01460225
Title: Effects of Lubiprostone on Gastric Sensory and Motor Function in Patients With Chronic Idiopathic Constipation
Brief Title: Effects of Lubiprostone on Gastric Function in Patients With Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 07-033L
Record Dates: First submitted 2010-07-19; First posted 2011-10-26 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Chronic Idiopathic Constipation
Keywords: constipation; chronic idiopathic constipation; no prior history of surgery to the colon; not on any type of medication that could alter gastrointestinal motility or transit
MeSH Terms: conditions — Constipation | interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): 24 micrograms of lubiprostone twice daily for one week.
  Interventions: Drug: lubiprostone

INTERVENTIONS:
Drug: lubiprostone — 24 micrograms twice daily for 1 week

SUMMARY:
This prospective study is designed to evaluate how lubiprostone may affect gastric motor and sensory function.

ELIGIBILITY:
Inclusion Criteria:

* chronic idiopathic constipation

Exclusion Criteria:

* medications that slow gastrointestinal (GI) motility
* prior surgery to the GI tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 patients entered the study; no dropouts. All patients completed the study; the entire study was contacted at Dartmouth.
Pre-assignment Details: No patients were excluded.
Period: Overall Study
Arm/Group | Lubirprostone
Started | 19 (January 2009.)
Completed | 19 (November 2010)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lubirprostone
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying
Description: gastric emptying was measured before and after 7 days of treatment.at set times (2 and 4 hours post eating a radio-labeled meal)
Time Frame: Day 1 and Day 7
Measure: Mean (Standard Deviation); unit: percent meal retention
Arm/Group | Prior to Treatement With Lubiprostone | Post Treatment With Lubiprostone
Number analyzed (Participants) | 19 | 19
percent meal retention
  2 Hours after meal | 0.27 (NA) — Original Data for this study have been destroyed, the study was not published and the Standard Deviation was not reported with the data in the only report available. A p= .003 was documented. This is the only measure of precision in the report. | 0.384 (NA) — Original Data for this study have been destroyed, the study was not published and the Standard Deviation was not reported with the data in the only report available. A p= .003 was documented. This is the only measure of precision in the report.
  4 Hours after meal | 0.04 (NA) — Original Data for this study have been destroyed, the study was not published and the Standard Deviation was not reported with the data in the only report available. A p value was documented and this is the only measure of precision in the report. | 0.051 (NA) — Original Data for this study have been destroyed, the study was not published and the Standard Deviation was not reported with the data in the only report available. A p value was documented and this is the only measure of precision in the report.
Statistical Analysis 1: Comparison: Prior to Treatement With Lubiprostone vs Post Treatment With Lubiprostone; Comparison of meal retention between pre-treatment and post treatment at 2 hours post meal; Test type: Equivalence — Based on the results of Camilleri et al, this should be adequate to detect up to a 30% difference in gastric emptying scan times with a p-value of 0.05 and 80% power; p = 0.003, t-test, 2 sided
Statistical Analysis 2: Comparison: Prior to Treatement With Lubiprostone vs Post Treatment With Lubiprostone; Comparison of meal retention between pre-treatment and post treatment at 4 hours post meal; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.122, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | All- Single Arm
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 2/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All- Single Arm (N=19)
nausea (Gastrointestinal disorders) | 2 (2) — 2 patients had nausea
Headache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No